CLINICAL TRIAL: NCT06773949
Title: Randomized Trial Assessing the Feasibility of Exercise as a Priming Strategy for rTMS Treatment in Difficult-to-Treat Depression
Brief Title: Feasibility Trial of Exercise as a Priming Strategy for rTMS Treatment in Difficult-to-Treat Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Sara Tremblay, Scientist, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0227
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD); Treatment Resistant Depression (TRD)
Keywords: iTBS; rTMS; Exercise; Physical inactivity
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 4-weeks of exercise (moderate-to-vigorous intensity) followed by 6 weeks of iTBS combined with exercise.
  Interventions: Device: Theta burst stimulation
- Standard Group (Other): Standard care of 4 weeks of stable treatment (i.e. no changes to antidepressant regimen or physical activity) followed by 6 weeks of iTBS alone.
  Interventions: Device: Theta burst stimulation

INTERVENTIONS:
Device: Theta burst stimulation — Cool B70 cooled-coil (left DLPFC) with X100 MagPro rTMS Device (Magventure A/S, Farum, Denmark)
  Other Names: rTMS

SUMMARY:
The goal of this study is to collect feasibility data on combining structured exercise aimed to improve physical fitness, and intermittent TBS (iTBS) in treating individuals diagnosed with difficult-to-treat depression who are physically inactive. By conducting this trial, we will compare the therapeutic benefits of the combined approach against the standard treatment of iTBS alone (without exercise). These findings will be used to inform future large-scale projects in which we will investigate, in a larger sample size, whether structured exercise aimed to improve fitness as recommended by most public exercise guidelines (i.e., ≥3x/week, moderate-to-vigorous intensity) serves as an active ingredient that amplifies the effectiveness of iTBS. Ultimately, the insights gained from this study will be valuable for clinicians seeking to alleviate depressive symptoms in MDD through neuromodulation techniques such as iTBS.

DETAILED DESCRIPTION:
This is a randomized, two-arm, pilot feasibility clinical trial design involving physically inactive individuals diagnosed with treatment-resistant depression (TRD). Participants will be randomly assigned to either: 1) 4-weeks of exercise (moderate-to-vigorous intensity; ~1h session, 3x/week) followed by 6 weeks of iTBS combined with exercise (intervention group), or 2) 4 weeks of stable treatment (i.e. no change in psychotropic medication/psychotherapy regimen or physical activity) followed by 6 weeks of iTBS alone (control group). The intervention group is divided into two phases: the priming phase and the synergetic phase. Due to the neuroplasticity-enhancing effects of exercise and fitness, and based on pilot results demonstrating superior antidepressant effects of TBS in physically active participants, the main objective of the priming phase is to enhance brain plasticity mechanisms through increases in fitness from the 4 weeks of exercise training. In other words, this phase aims to build capacity for a better response to TBS treatment. The synergetic phase (interventional group) follows the priming and involves integrating TBS treatment into the exercise training regimen. Participants in the interventional group will maintain their exercise routine to enhance and sustain gains while undergoing TBS treatment for 6 weeks. In accordance with the recommended guidelines for both exercise and TBS treatment for depression, participants in the interventional group will engage in exercise sessions lasting approximately 1 hour, three times per week. In both interventional and control groups, TBS treatment will be administered five times per week, with treatment delivery lasting 3 minutes. We hypothesize that all aspects of this project will be feasible, that is the exercise and iTBS delivery and outcomes assessment. Additionally, we expect participants to show high levels of adherence and compliance with the strategy. The ultimate goal, to be investigated in a larger-scale study following this one, is to determine whether exercise acts as an active ingredient that enhances the effectiveness of iTBS.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 18-75 years old.
2. Able to provide voluntary informed consent.
3. Diagnosis of MDD or Persistent Depressive Disorder, without psychotic features, confirmed by MINI for DSM-5.
4. Depressive symptoms have not improved after ≥ 1 adequate antidepressant trial in the current episode (i.e., difficult-to-treat MDD), based on the Antidepressant Treatment History Form (ATHF).
5. Baseline score of ≥15 on the HRSD-17.
6. No change in psychotropic medications or psychotherapy regimen at least 4 weeks prior to entering the trial
7. Physically inactive as per the International Physical Activity Questionnaire - Short Form (IPAQ-SF).
8. Able to engage in structured exercise as per the Get Active Questionnaire (GAQ).
9. Able to adhere to the proposed treatment schedule.

Exclusion Criteria:

1. Diagnosis of bipolar I or II disorder, based on DSM-5 criteria.
2. Current or past (<3 months) substance (excluding caffeine or nicotine) or alcohol abuse/dependence, as defined in DSM-5 criteria.
3. Current use of illegal substances.
4. Current use of cannabis.
5. Concomitant major unstable medical or neurologic illness (e.g., uncontrolled diabetes or renal dysfunction).
6. Organic cause of the depressive symptoms (e.g. thyroid dysfunctions), determined by the referring physician.
7. Acute suicidality or threat to life from self-neglect.
8. Pregnant or breastfeeding, or thinking of becoming pregnant during course of treatment.
9. Contraindication for TMS and MRI (e.g., personal history of epilepsy or seizure, metallic head implant, pacemaker), confirmed by TMS Adult Safety Scale (TASS) and MRI pre-screener.
10. Unwilling to maintain current psychotropic medication and/or psychotherapy regimen for the four weeks prior to and for the duration of the study.
11. Taking more than 1 mg/day of lorazepam or equivalent.
12. Any other condition that, in the opinion of the investigators which would adversely affect the participant's ability to complete the study.
13. Physically active: performing exercise and/or physical activity levels meeting the cut-off for "minimally active" on the IPAQ-SF.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Assessing feasibility on combining structured exercise and intermittent Theta Burst Stimulation (iTBS) in participants with treatment-resistant depression (TRD) | Assessed at the end of the study once all participants have completed the study.
  Feasibility outcomes are crucial metrics that will guide the refinement of our protocols, thereby enhancing our preparedness for future design endeavors. These will include: 1) recruitment, 2) adherence, 3) compliance, 4) retention, 5) satisfaction, and 6) adverse events.
Compare the effects on clinical response of exercise on enhancing iTBS treatment efficacy vs. iTBS alone | Administered at screening, before iTBS treatment course (week 4), at the end of the treatment course (week 10), then at the 6-week follow-up (week 16)
  Clinical response will be defined as a ≥ 50% reduction in the 17-item Grid Hamilton Rating Scale for Depression (Grid-HRSD-17). The Grid HRSD is a clinician-rated instrument with seventeen items used to measure the severity of depressive episodes. The overall score ranges from 0 to 52, where scores of 0 to 7 are considered as being normal, 8 to 16 suggest mild depression, 17 to 23 moderate depression, and scores ≥ 24 indicate severe depression.

SECONDARY OUTCOMES:
Change in self-reported depression symptoms as measured by Beck Depression Inventory (BDI-II). | Administered at screening, before the first iTBS treatment (week 4) and every week after that for 6 weeks (week 5, week 6, week 7, week 8, week 9, week 10), and at the 6-week follow-up assessment (week 16)
  As a secondary measure of depressive symptoms. Score scale from 0 (better outcome, no depression) to 63 (worst outcome, extreme depression).
Change in self-reported anxiety symptoms as measured by Beck Anxiety Inventory (BAI) | Administered at screening, before the first iTBS treatment (week 4) and every week after that for 6 weeks (week 5, week 6, week 7, week 8, week 9, week 10), and at the 6-week follow-up assessment (week 16)
  As a secondary measure of anxiety symptoms. Score scale from 0 (better outcome, no depression) to 63 (worst outcome, extreme anxiety).
Change in self-reported suicidal thoughts symptoms as measured by Beck Scale for Suicidal Ideation (BSS) | Administered at screening, before the first iTBS treatment (week 4) and every week after that for 6 weeks (week 5, week 6, week 7, week 8, week 9, week 10), and at the 6-week follow-up assessment (week 16)
  To assess the effect of treatment on suicidal thoughts that may be improved by iTBS.
  Score scale from 0 (better outcome, no desire for suicide) to 38 (worst outcome, extreme desire for suicide).
Change in self-reported hopelessness as measured by State Hope Scale (SHS) | Administered at screening, before the first iTBS treatment (week 4) and every week after that for 6 weeks (week 5, week 6, week 7, week 8, week 9, week 10), and at the 6-week follow-up assessment (week 16)
  To assess the effect of treatment on self-report symptoms and perceptions of stress that may be improved by iTBS.
  6-item measure where responses are rated on an 8-point Likert scale. Score scale from 1 (Definitely True) to 8 (Definitely False).
Change in neuroplasticity as measured by neurophysiology (TMS) and MRI (Arterial Spin Labelling measures of brain blood flow) | Administered at pre-assessment (baseline), before iTBS treatment course (week 4), end of iTBS treatment course (week 10)
  To assess the effect of treatment on biomarkers. Greater improvements in these biomarkers will also be associated with greater reductions in depressive symptoms.
Change in grip strength as measured by dynamometer | Administered at pre-assessment (baseline), before iTBS treatment course (week 4), end of iTBS treatment course (week 10), and at 6-week follow-up assessment (week 16)
  To assess the effect of treatment on biomarkers. Greater improvements in these biomarkers will also be associated with greater reductions in depressive symptoms.
Change in physical measures as assessed by anthropometrics | Administered at pre-assessment (baseline), before iTBS treatment course (week 4), end of iTBS treatment course (week 10), and at 6-week follow-up assessment (week 16)
  To assess the effect of the intervention on physical health.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (16 weeks).
  Adverse events will be tracked and recorded.
Side Effects | Daily Monday-Friday throughout study (16 weeks).
  Side effects will be tracked and recorded on any TMS visits, using the TMS side effects questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tremblay, PhD, Principal Investigator — Royal Ottawa Mental Health Centre
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data collected from this study (IPD) will be de-identified for all parties who have permission to access it. This de-identified data may be shared with other researchers at the Royal's Institute of Mental Health Research. De-identified may be shared with the public only upon request. Please note that all data that has the potential of revealing participants' identity will NOT be used to share.
Time Frame: De-identified data may become available (upon request) when the study is completed and published (anticipated time frame: the year of 2027)
Access Criteria: De-identified data will be accessible only through the permission of the lead research scientist. All requests must be made and accepted by her.